CLINICAL TRIAL: NCT00783393
Title: SCH 52365 Phase II Clinical Study: A Study on the Efficacy and Safety of Monotherapy With SCH 52365 in Patients With First Relapsed Anaplastic Astrocytoma
Brief Title: SCH 52365 Phase II Clinical Study: A Study on the Efficacy and Safety of Monotherapy With SCH 52365 in Patients With First Relapsed Anaplastic Astrocytoma (Study P03745)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03745; JPC02-351-21
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Astrocytoma
MeSH Terms: conditions — Astrocytoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): The study consists of two steps:
  * Step 1, the therapeutic study phase, comprising six cycles of treatment with temozolomide, and
  * Step 2, the long-term treatment phase, where subjects with at least disease stabilization at the end of Step 1 may continue temozolomide treatment until unacceptable toxicity or disease progression occur, up to a maximum of 2 years from the start of treatment in Cycle 1.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide orally once daily for 5 consecutive days followed by a 23 day rest period to complete a 28 day treatment cycle. In Cycle 1, temozolomide will be administered at 150 mg/m2/day; in Cycle 2 and subsequent cycles, it will be administered at 100, 150, or 200 mg/m2, depending on hematology test results and adverse events observed.
  Other Names: Temodal, Temodar, SCH 052365

SUMMARY:
The primary purpose of the study is to evaluate the efficacy (overall response) and safety of temozolomide in Step 1 at the dose and regimen approved in the US and the EU countries (28 day cycles of temozolomide at 150 to 200 mg/m2 once daily for 5 consecutive days with a 23 day rest period) in patients with anaplastic astrocytoma at first relapse.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically confirmed anaplastic astrocytoma on the tentorium at first relapse, and satisfy the following:

  * unequivocal evidence of tumor recurrence or aggravation by MRI scan after treatment for initial onset; the lesions must be measurable;
  * anaplastic astrocytoma diagnosed histologically by the last pathological diagnostic tests (including initial diagnosis) prior to initial administration of temozolomide;
  * tissue samples available for Central Pathologic Reviewer;
  * pathologic diagnosis report by the study-conducting medical institution must be available for the sponsor.
* MRI-related criteria:

  * MRI scan performed within 14 days before initial temozolomide administration;
  * assessable tumor site confirmed by MRI;
  * dosage of steroidal agents not increased within 7 days before MRI prior to initial temozolomide administration, except for postoperative subjects for first relapse;
  * MRI performed at the Principal Investigator's study location or designated radiology facility during the study.
* Age >=18 years, either sex, inpatients or outpatients.
* Use of medically approved contraception methods in fertile subjects.
* Karnofsky performance status >=70.
* Adequate clinically laboratory values obtained within 14 days before initial temozolomide administration.
* Criteria regarding treatment of initial onset:

  * tumor biopsy, regardless of tumor resection at initial diagnosis;
  * prior radiation therapy;
  * prior chemotherapy with up to one nitrosourea-containing regimen.
* Tumor may or may not have been surgically resected at first relapse, but residual measurable disease is required.
* For subjects who had surgical resection of tumor at first relapse:

  * MRI scan must have been performed within 72 hours after surgery.
  * the dose of steroidal agents must be reduced before temozolomide administration.
* Life expectancy >=12 weeks.
* Written informed consent obtained.

Exclusion Criteria:

* History of treatment with dacarbazine.
* Subjects who received chemotherapy within 6 weeks before initial temozolomide administration.
* Subjects who received interstitial radiotherapy or stereotactic radiosurgery.
* Subjects who completed radiotherapy within 12 weeks before initial temozolomide administration.
* Surgery at first relapse (including biopsy) within 1 week before initial temozolomide administration.
* Subjects not recovered from acute toxicity due to previous therapy.
* High-risk subjects with complication of diseases other than malignant tumor, or who require systemic administration of antibiotics for infection.
* Previous or concurrent malignancies at other sites.
* Pregnant or nursing women.
* Women of childbearing potential not using an effective method of contraception.
* Subjects previously treated with temozolomide.
* Participation in an ongoing clinical study, or in other clinical studies within 6 months before initial temozolomide administration.
* Subjects found inappropriate for the study by the investigator or subinvestigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-05-27 (Actual); Primary Completion 2005-06-17 (Actual); Study Completion 2005-06-17 (Actual)

PRIMARY OUTCOMES:
Overall response in Step 1 | 6 months
Incidence rate and severity of adverse events with administration of temozolomide in Step 1 | 7 months (during temozolomide administration for 6 months and follow-up for 1 month)

SECONDARY OUTCOMES:
Progression-free survival in Step 1 | 6 months
Overall survival in Step 1 | 6 months
Tumor response in Step 1 | 6 months
Neurological improvement in Step 1 | 6 months
Progression-free survival, overall survival, overall response, effect on neurological symptoms, and safety in Step 2 | 6 months
Progression-free survival in Step 2 | Up to 2 years
Overall survival in Step 2 | Up to 2 years
Overall response in Step 2 | Up to 2 years
Effect on neurological symptoms in Step 2 | Up to 2 years
Safety in Step 2 | Up to 2 years

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html